CLINICAL TRIAL: NCT02828397
Title: A Randomized, Open-Label, Parallel Group Study of the Pharmacokinetics, Safety, and Tolerability of a Single Intramuscular (IM) Injection of REGN2222 Produced by 2 Different Cell Lines in Healthy Adult Subjects
Brief Title: Study of the Blood Concentrations of Two Formulations of REGN2222 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: R2222-HV-1520
Record Dates: First submitted 2016-07-07; First posted 2016-07-11 (Estimated); Last update posted 2016-11-04 (Estimated); Status verified 2016-11

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Reference Drug (Experimental): REGN2222 Reference Formulation
  Interventions: Drug: REGN2222
- Test Drug (Experimental): REGN2222 Test Formulation
  Interventions: Drug: REGN2222

INTERVENTIONS:
Drug: REGN2222

SUMMARY:
Primary Objective: Determine blood concentrations of two formulations of REGN2222

Secondary Objective: Assess safety and tolerability of REGN2222

ELIGIBILITY:
Key Inclusion Criteria:

1. Healthy man or woman aged 18 to 60 years
2. Body weight between 50.0 kg and 95.0 kg, inclusive
3. Willing and able to comply with clinic visits and study-related procedures
4. Provide signed informed consent

Key Exclusion Criteria:

1. Hemoglobin not within normal limits
2. Positive drug and alcohol screen test results at screening visits 1 and 2
3. Participation in any clinical research study that evaluated another investigational drug or therapy within 30 days or at least 5 half-lives, whichever is longer, of the investigational drug, prior to the screening visit
4. Pregnant or breastfeeding women, and women of childbearing potential
5. Sexually active men who are unwilling to practice adequate contraception during the study

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2016-04; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Serum REGN2222 concentration-time curve (AUC) | Day 1 to Day 148 (end of study)
Peak REGN2222 concentration (Cmax) | Day 1 to Day 148 (end of study)

SECONDARY OUTCOMES:
Treatment-emergent adverse events (TEAEs) from baseline to the end of the study | Day 1 to Day 148 (end of study)
Presence or absence of anti-drug antibody (ADA) | Day 1 to Day 148 (end of study)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Management, Study Director — Regeneron Pharmaceuticals
Locations (2):
- United States (2):
  - Daytona Beach, Florida
  - Evansville, Indiana